CLINICAL TRIAL: NCT02669654
Title: Effectiveness Trial of Day-care Versus Usual Care Management of Severe Pneumonia With or Without Malnutrition in Children Using the Existing Health System of Bangladesh
Brief Title: Effectiveness Trial of Day-care vs. Usual Care of Severe Pneumonia & Malnutrition in Children
Acronym: Day-care
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: UBS Optimus Foundation (Other); UNICEF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-14066
Record Dates: First submitted 2015-12-01; First posted 2016-02-01 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-02

CONDITIONS: Pneumonia Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Day-care management of Severe Pneumonia (Experimental): management in Day-care clinic
  Interventions: Other: Day-care management of Severe Pneumonia
- Existing Treatment Centre (ETC) (No Intervention): Severe Pneumonia management in Existing Treatment Centre

INTERVENTIONS:
Other: Day-care management of Severe Pneumonia — Day-care management of Severe Pneumonia
  Arms: Day-care management of Severe Pneumonia

SUMMARY:
Background: At present pneumonia and malnutrition have become the leading causes of mortality among <5-year-old children in developing countries. World Health Organization standard management of severe pneumonia and severe malnutrition requires hospitalization for supportive care. As many developing countries including Bangladesh do not have enough pediatric hospital beds to accommodate the demand for admission of all children with severe pneumonia and malnutrition, Investigators developed alternative treatment option such as "Day Care Approach", for those children who cannot be hospitalized, but are too sick to be managed in the community. After successful Day Care Approach of management of efficacy trials with severe childhood pneumonia and severe malnutrition, the next step is to conduct an effectiveness trial under "real life" condition, i.e. within the Health Systems of Bangladesh.

Burden: Pneumonia is the leading cause of mortality in developing countries, being responsible for 1,368,000 (18%) of annual 7.6 million deaths, 95% occurring in developing countries. Similarly, malnutrition is a major health problem with an estimated 1.7 & 3.6 million children dying annually because of Severe Acute Malnutrition & Moderate Acute Malnutrition, respectively.

Objectives: To assess & implement the Day Care Approach of management of severe childhood pneumonia with or without Moderate Acute Malnutrition and/or severe underweight into existing Health Systems of Bangladesh as a safe & cost effective alternative to Existing Treatment.

Methods: A cluster randomized controlled trial will be conducted in Bangladesh by involving 16 clusters (Wards) in Dhaka & 16 clusters (Unions) in rural areas that will be randomly assigned to intervention & control arm. Children with severe pneumonia will be enrolled in (i) Tikatuli, (ii) Circular Road, (iii) Dhamrai Upazilla of Dhaka, (iv) Karimganj Upazillas to one of two management schemes: (i) Existing Treatment in control clusters or (ii) Day care Approach in intervention clusters by involving Comprehensive Reproductive Health Centres in urban and Health and Family Welfare Centres in rural areas.

Outcome variables:

* Primary: clinical treatment failure by day 6
* Secondary:

  (i) Treatment failure between day 7-14 in children who are well on day 6 (ii) Cost effectiveness (iii) Referrals to hospitals (iv) Deaths

DETAILED DESCRIPTION:
Specific Objectives:

1. To assess whether or not the Day care Approach for the management of severe childhood pneumonia with or without moderate acute malnutrition and/or severe underweight incorporated into the existing urban and rural Health Systems of Bangladesh is safe and effective.
2. To implement the Day care Approach for the management of severe childhood pneumonia with or without moderate acute malnutrition and/or underweight within the Health Systems of Bangladesh as a cost effective alternative to the Existing Treatment of care for both the Health Systems and the families.
3. To examine and compare the cost effectiveness of the Day care Approach versus Existing Treatment of care for the management of severe childhood pneumonia with or without moderate acute malnutrition and/or severe underweight.
4. To identify and assess potential barriers and challenges during the whole implementation process.

Background of the Project including Preliminary Observations:

At present and depending on clinical presentation, pneumonia is classified as severe pneumonia, pneumonia, or no pneumonia, according to the recent guidelines by the World Health Organization in 2013. Since pneumonia is the leading cause of death in <5-year-old children, interventions to promote the prevention and treatment of pneumonia are an essential part of child survival efforts to achieve Millennium Development Goal 4. World Health Organization standard management of severe pneumonia requires hospitalization for supportive treatment including oxygen therapy for hypoxaemia, airway suctioning, fluid and nutritional management, antibiotics, and careful monitoring.

Most, if not all, developing countries including Bangladesh do not have enough hospitals, or pediatric hospital beds to accommodate the demand for admission of all children with severe pneumonia with or without malnutrition and other co-morbidity. In addition, mothers of ill children have other childcare and household responsibilities that constrain their ability to attend the child during hospitalization, which is often mandatory. Furthermore, transportation, cost, long distance from the hospital, lack of adequate child-care at home, or cultural perceptions represent additional huge limitations to hospitalization. Hospitalization also may not be feasible due to inability of parents to stay in hospital for the entire duration of illness. The sum total of all these common potential constraints lead to failure of hospitalization of children with severe pneumonia and severe malnutrition with or without additional co-morbidity. This inadequate availability and use of hospital beds leading to failure of hospitalization of children with severe pneumonia and/or malnutrition assuredly results in excess and unwanted deaths of children, who, with proper care, would otherwise survive. Although Investigators do not have direct evidence (no data available) that the bottleneck to pneumonia deaths in Bangladesh is lack of hospital beds mainly. But Investigators know from experience that many children with severe pneumonia requiring hospitalization are not hospitalized due to the lack of free pediatric beds, as observed during the observational day care studies.

Study Design A cluster randomized controlled clinical trial will be conducted in urban Dhaka and rural Bangladesh. The trial areas are pre-selected on the basis of infrastructure (adequate space, water supply, electricity, and willingness for performing the study). In the urban areas, 16 clusters equivalent to Wards (either whole or partial), with a population of 50,000 to 80,000 each and in the rural areas, another 16 clusters equivalent to Unions each with about 20,000 to 30,000 inhabitants. Children with severe pneumonia, according to recent World Health Organization criteria (2013) with or without malnutrition will be enrolled into the study in urban Dhaka: (i) Tikatuli, Surjer Hashi Clinic, 12, K.M. Das Lane and (ii) Circular Road Circular Road Surjer Hashi Clinic, New Circular Road; and rural Bangladesh: (iii) Dhamrai Upazilla of Dhaka District, and (iv) Karimganj Upazilla of Kishoreganj District to one of the two management schemes: (i) the Existing Treatment in the control clusters, or (ii) the Day care Approach in the intervention clusters. Children with history of cough, fever and difficult breathing suggestive of having severe pneumonia will be enrolled at primary health facilities such as Primary Health Care Centres or Comprehensive Reproductive Health Centres in the urban areas and Health and Family Welfare Centres or Community Clinics in the rural areas.

Methods

Primary study sites Urban: United States Agency for International Development -Department For International Development support Non Government Organization Health Service Delivery Project through Pathfinder run by the Population Services and Training Center and Concerned Women for Family Development. The Ministry of Health and Family Welfare contributes to urban health care through the outpatient services offered through its secondary, tertiary and specialized hospitals located in the urban settings.

Rural: Health services in Bangladesh in the rural areas are mostly provided by the Government's Ministry of Health and Family Welfare, Non-Government Organizations (NGOs), and private providers. In the government sector, two community based workers - a family welfare assistant and a health assistant - and a community clinic run by a community health care provider serve a population of 6000 to 7000. Another first level outpatient clinic - e.g. Union Health and Family Welfare Centres - serves a population of about 20,000.

Randomization and masking The trial field sites have been pre-selected on the basis of infrastructure (adequate space, water supply, electricity and willingness for performing the study).

Case Management

Existing Treatment (control) clusters

Children in the control Existing Treatment clusters with pneumonia (not severe pneumonia) with/without malnutrition will be identified by the Community Health Worker/Community Service Providers in the urban areas or Field Research Assistants/Field Assistants in the rural areas, or self-referred by the parents/caregivers to the Primary Health Care Centres (Vital clinics)/Comprehensive Reproductive Health Centres (Ultra clinics) in the urban areas and Community Clinics/Health and Family Welfare Centres in the rural areas.

Follow-up in the Existing Treatment control clusters

Community Health Workers/Field Research Assistants/Field Assistants will perform the follow-up visits at the clinics on days 2, child's home on day 3, and clinics on day 6 and day 14 (window period + 1 day) in the Existing Treatment clusters of all four primary study sites.

In case of treatment failure in control areas children will be referred to hospital from Day 2.

Day Care Approach (Intervention) clusters

Similarly, children of the intervention Day care Approach clusters with pneumonia (not severe pneumonia) with or without malnutrition will be addressed in the same manner as the control clusters, i.e. be identified by the Community Health Workers in the urban areas and Field Research Assistants/Field Assistants in the rural areas. As with the children in the control clusters at the 1st level care centres (Primary Health Care Centres/Comprehensive Reproductive Health Centres in the urban areas and Community Clinics/Health and Family Welfare Centres in the rural areas), the children will be assessed by the Physicians/Pediatricians working at the Comprehensive Reproductive Health Centres in the urban areas and by the Sub Assistant Community Medical Officers working at the Health and Family Welfare Centres in the rural areas and finally evaluated by a trained study physician and treated at home with oral antibiotics (syrup Amoxicillin 90 mg/kg three divided doses or Co-trimoxazole 40 mg/kg two divided doses per day for 5 days).

Children with pneumonia (i.e., not severe pneumonia) who fail to the community level oral Amoxicillin/Co-trimoxazole treatment for two days as well as those presenting with severe pneumonia (self-referred or identified by Community Health Workers/Field Research Assistants/Field Assistants) right from beginning will be assessed by the Physicians/Pediatricians working at the Comprehensive Reproductive Health Centres in the urban areas and by the Sub Assistant Community Medical Officers working at the Health and Family Welfare Centres in the rural areas and finally evaluated by a trained study physician and directly referred to the Comprehensive Reproductive Health Centres in the urban areas or Health and Family Welfare Centres in the rural areas for Day care Approach of management. For this purpose, the children will be admitted to a day-care section of the Comprehensive Reproductive Health Centres in the urban areas from 08:30 to 17:00 hours and to a day-care section of the Health and Family Welfare Centres in the rural areas from 08:30 to 15:00 hours on all days of the week including weekends and public holidays, until fulfilling the criteria for discharge (clinical end-points, defined as no hypoxemia, no fever, no fast breathing and no tachycardia). Parents will bring their children to the Comprehensive Reproductive Health Centres/Health and Family Welfare Centres at 8:30 hours in the morning every day and return them back home at 15:00 hours in rural areas or 17:00 hours in urban areas.

Follow-up study up to 3 months after discharge

After successful management of all enrolled study children belonging to all Existing Treatment/Day care Approach clusters will be discharged from the Comprehensive Reproductive Health Centres/Health and Family Welfare Centres. The study physicians will inform the parents on the dates of follow-up visits for the next 3 months written down in the discharge certificate.

Economic Evaluation of Intervention Alternatives

Effectiveness trial of severe pneumonia without/with Moderate Acute Malnutrition and or severe underweight is planned to implement the Day care Approach of treatment into the urban Comprehensive Reproductive Health Centres in Dhaka city or the rural Health and Family Welfare Centres of Bangladesh.

Cost of intervention

Intervention costs consist of the costs of providers and households.

Cost of provider Cost to household

Sample Size Calculation and Outcome (Primary and Secondary) Variable(s)

Cluster-randomized design for dichotomous outcomes with an equivalency design and the explicit expectation that the results on primary outcomes would fall within the 95% Confidence Intervals. Because the number of clusters is fixed at 8 clusters per site per year including 4 control and 4 intervention and a power of 90%, coefficient of variation of 0.20, and an alpha of 0.05. On the basis of these assumptions, 50 children with severe pneumonia with or without malnutrition with or without severe under-weight per cluster per year will be enrolled over 2.5 years, for an estimated 2000 patients in each study arm including 15% drop-outs. 32 clusters will be needed in each study arm. Therefore, for a period of 2.5 years, a total of 4000 children can be easily recruited within the time frame from 4 primary study sites. The estimated incidence of pneumonia is taken as 0.23 episode/ child/ year.

Outcome Variables

* The primary outcome variable will be the following (i) Clinical treatment failure by day 6 after enrollment (ii) Success rate of the Health System Day acre Approach plus referral to hospital verses Existing Treatment plus referral to hospital)
* The secondary outcome variables will be:

(iii) Treatment failure or relapse between day 7 and day 14 in children who are well on day 6 (iv) Economic evaluation (cost-effective analyses) (v) Referrals to hospitals (vi) Deaths (vii) Compliance to treatment (viii) Anthropometrical indices such as body weight, length/height, Mid Upper Arm Circumference, Weight-for-Age (%), Weight-for-Height (%), Height-for-Age (%) (ix) Morbidity, mortality, relapse and hospitalization during 3-months follow-up after discharge from the study (x) Family/patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* 2 to 59 months of age
* Both male and female
* Severe pneumonia with at least one of the following signs:
* Central cyanosis
* Hypoxaemia (Oxygen saturation < 90% on pulse oximetry)
* Severe respiratory distress
* Grunting
* Very severe chest indrawing
* Signs of pneumonia with a general danger sign
* Inability to breastfeed or drink
* Lethargy
* Reduced level of consciousness
* Unconsciousness
* Convulsions
* Severe pneumonia with associated illnesses such as the following:
* Moderate Acute Malnutrition
* Severe under-weight [Weight-for-Age Z-score <-3]
* Diarrhea with no or some dehydration
* Living in the study area (in one of the above four primary study sites)
* Informed consent given by parents/legal guardian

Exclusion Criteria:

* Pneumonia
* No pneumonia
* Hospital-acquired/nosocomial pneumonia
* Bronchiolitis
* Severe Acute Malnutrition
* Associated other severe diseases of childhood such as:
* diarrhea with severe dehydration
* Shock/severe sepsis
* Meningitis/encephalitis
* Bronchial asthma
* Congenital Heart Disease
* Participated in this study once and other study in the past 2 weeks
* Received parenteral antibiotics for the current illness
* Parents or legal guardians refusal to participate

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical treatment failure by day 6 from severe pneumonia in the Day care clinics compare to the patients who will get treatment from Hospitals | 6 days
  Patients will not recover within day 6 from severe pneumonia in the Day care clinics

SECONDARY OUTCOMES:
Treatment failure between day 7-14 in children who are well on day 6 from severe pneumonia in the Day care clinics compare to the patients who will get treatment from Hospitals | 14 days
  Patients will recover within day 6 from severe pneumonia in the Day care clinics but again will have severe pneumonia within day 7-14

CONTACTS AND LOCATIONS:
Overall Officials: Nurul Hoque Alam, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (2):
- Bangladesh (2):
  - Icddr,B, Dhaka
  - Rural and Urban areas in Bangladesh, Dhaka

REFERENCES:
- [Derived] Alam NH, Faruque AS, Ashraf H, Chisti MJ, Ahmed T, Sultana M, Khalequzzaman M, Ali S, Ahmed S, Nasrin S, Tariqujjaman M, Huq KATME, Amin R, Mollah AH, Kabir L, Shahidullah M, Khanam W, Islam K, Kim M, Vandenent M, Duke T, Gyr N, Fuchs GJ. Effectiveness, safety and economic viability of daycare versus usual hospital care management of severe pneumonia with or without malnutrition in children using the existing health system of Bangladesh: a cluster randomised controlled trial. EClinicalMedicine. 2023 Jun 6;60:102023. doi: 10.1016/j.eclinm.2023.102023. eCollection 2023 Jun. PMID 37304498